CLINICAL TRIAL: NCT07078318
Title: The Effect of Respiratory Exercises Given in Addition to Pelvic Floor Rehabilitation on Dyspareunia and Autonomic Nervous System in Women With Musculoskeletal Dyspareunia
Brief Title: Effect of Respiratory Exercises With Pelvic Floor Rehab on Dyspareunia & Autonomic Function in Women
Acronym: Dyspareunia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya Applied Sciences University (Other)
Responsible Party: Principal Investigator, Abdurrahim Yıldız, Assoc. Prof., Sakarya Applied Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2025-07-03; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Dyspareunia (Female Excluding Psychogenic); Female Sexual Dysfunction (FSD); Chronic Pelvic Pain
Keywords: Dyspareunia; Pelvic Floor Rehab; Manual Therapy; Autonomic Regulation; Sexual Dysfunction
MeSH Terms: conditions — Dyspareunia; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: A total of 45 participants aged 18-45 years who meet the inclusion criteria will be randomly assigned into three equal groups (n = 15):
  Group I: Pelvic floor rehabilitation only
  Group II: Pelvic floor rehabilitation + diaphragmatic breathing exercises
  Group III: Pelvic floor rehabilitation + diaphragmatic breathing exercises + diaphragm manual therapy
  Interventions will be administered once per week for 8 weeks. Pre- and post-intervention assessments will include pain intensity (Visual Analog Scale), pelvic floor muscle function (ultrasonography), sexual function (Female Sexual Function Index), anxiety level (Beck Anxiety Inventory), and autonomic regulation (Heart Rate Variability using Elite HRV).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: Pelvic floor rehabilitation (Experimental): Pelvic floor rehabilitation only
  Interventions: Other: Pelvic floor rehabilitation; Other: Diaphragmatic Breathing Exercises; Other: Diaphragm Manual Therapy
- Group II: Pelvic floor rehabilitation + diaphragmatic breathing exercises (Experimental): Pelvic floor rehabilitation + diaphragmatic breathing exercises
  Interventions: Other: Diaphragmatic Breathing Exercises; Other: Diaphragm Manual Therapy
- Group III: Pelvic floor rehabilitation + diaphragmatic breathing exercises + diaphragm manual therap (Experimental): Pelvic floor rehabilitation + diaphragmatic breathing exercises + diaphragm manual therapy
  Interventions: Other: Diaphragm Manual Therapy

INTERVENTIONS:
Other: Pelvic floor rehabilitation — Participants in this group will receive standard pelvic floor rehabilitation. This includes education about pelvic floor anatomy and function, supervised pelvic floor muscle training (Kegel exercises), relaxation techniques, and manual release of trigger points if necessary. The aim is to improve muscle strength, coordination, and reduce pelvic floor hypertonicity contributing to dyspareunia.
  Arms: Group I: Pelvic floor rehabilitation
Other: Diaphragmatic Breathing Exercises — In addition to the standard pelvic floor rehabilitation, participants in this group will practice diaphragmatic breathing exercises. These exercises focus on deep, slow nasal inhalation using the diaphragm, encouraging abdominal expansion while minimizing chest movement. Sessions are performed twice daily for 10 minutes. This technique is aimed at promoting parasympathetic activation, reducing anxiety, and improving autonomic regulation.
  Arms: Group I: Pelvic floor rehabilitation; Group II: Pelvic floor rehabilitation + diaphragmatic breathing exercises
Other: Diaphragm Manual Therapy — an additional manual therapy intervention targeting the diaphragm. Diaphragm manual therapy involves hands-on techniques applied to the thoracic and abdominal regions to reduce fascial restrictions, improve diaphragmatic mobility, and support deeper, more effective breathing. The therapy is delivered for 15 minutes at the start of each weekly session by a trained physiotherapist.

SUMMARY:
Background and Aim:

Dyspareunia, or pain during sexual intercourse, is a common component of female sexual dysfunction and may have multifactorial origins, including musculoskeletal and autonomic factors. While pelvic floor rehabilitation is an established treatment approach for musculoskeletal dyspareunia, it may not sufficiently address the autonomic dysregulation commonly observed in chronic pain conditions. The aim of this study is to investigate the effects of adding diaphragmatic breathing exercises and diaphragm manual therapy to standard pelvic floor rehabilitation on pain severity, pelvic floor function, and autonomic nervous system regulation in women diagnosed with musculoskeletal-origin dyspareunia.

Methods:

This randomized controlled clinical trial will be conducted between September 1, 2025, and December 1, 2025, at the Kurbaa Training and Consultation Center in Istanbul. A total of 45 participants aged 18-45 years who meet the inclusion criteria will be randomly assigned into three equal groups (n = 15):

Group I: Pelvic floor rehabilitation only

Group II: Pelvic floor rehabilitation + diaphragmatic breathing exercises

Group III: Pelvic floor rehabilitation + diaphragmatic breathing exercises + diaphragm manual therapy

Interventions will be administered once per week for 8 weeks. Pre- and post-intervention assessments will include pain intensity (Visual Analog Scale), pelvic floor muscle function (ultrasonography), sexual function (Female Sexual Function Index), anxiety level (Beck Anxiety Inventory), and autonomic regulation (Heart Rate Variability using Elite HRV). Statistical analyses will be performed using SPSS with significance set at p < 0.05.

Expected Contribution:

This study is expected to contribute to the development of more comprehensive treatment protocols for dyspareunia by integrating physical and neurophysiological rehabilitation components. It may also provide evidence supporting the role of autonomic regulation in improving treatment outcomes for female sexual pain disorders.

DETAILED DESCRIPTION:
Background and Aim:

Dyspareunia, or pain during sexual intercourse, is a common component of female sexual dysfunction and may have multifactorial origins, including musculoskeletal and autonomic factors. While pelvic floor rehabilitation is an established treatment approach for musculoskeletal dyspareunia, it may not sufficiently address the autonomic dysregulation commonly observed in chronic pain conditions. The aim of this study is to investigate the effects of adding diaphragmatic breathing exercises and diaphragm manual therapy to standard pelvic floor rehabilitation on pain severity, pelvic floor function, and autonomic nervous system regulation in women diagnosed with musculoskeletal-origin dyspareunia.

Methods:

This randomized controlled clinical trial will be conducted between September 1, 2025, and December 1, 2025, at the Kurbaa Training and Consultation Center in Istanbul. A total of 45 participants aged 18-45 years who meet the inclusion criteria will be randomly assigned into three equal groups (n = 15):

Group I: Pelvic floor rehabilitation only

Group II: Pelvic floor rehabilitation + diaphragmatic breathing exercises

Group III: Pelvic floor rehabilitation + diaphragmatic breathing exercises + diaphragm manual therapy

Interventions will be administered once per week for 8 weeks. Pre- and post-intervention assessments will include pain intensity (Visual Analog Scale), pelvic floor muscle function (ultrasonography), sexual function (Female Sexual Function Index), anxiety level (Beck Anxiety Inventory), and autonomic regulation (Heart Rate Variability using Elite HRV). Statistical analyses will be performed using SPSS with significance set at p < 0.05.

Expected Contribution:

This study is expected to contribute to the development of more comprehensive treatment protocols for dyspareunia by integrating physical and neurophysiological rehabilitation components. It may also provide evidence supporting the role of autonomic regulation in improving treatment outcomes for female sexual pain disorders.

ELIGIBILITY:
Inclusion Criteria:

Female participants aged between 18 and 45 years

Experiencing dyspareunia of musculoskeletal origin for at least 6 months

In a stable sexual relationship and sexually active

Willing and able to attend weekly treatment sessions for 8 weeks

Able to provide informed consent

No pelvic surgery within the last 6 months

Normal cognitive function and ability to follow instructions

Baseline FSFI score indicating sexual dysfunction (e.g., ≤ 26.55)

Exclusion Criteria:

* Presence of neurological, gynecological, or urological pathologies causing pelvic pain (e.g., endometriosis, pelvic inflammatory disease)

Pregnancy or postpartum period within the last 6 months

Diagnosed psychiatric disorders (e.g., major depression, psychosis)

Use of medications that affect autonomic nervous system function (e.g., beta-blockers, antidepressants)

History of pelvic radiation, cancer, or pelvic trauma

Participation in other rehabilitation or psychotherapy programs during the study period

Inability to tolerate manual therapy or perform breathing exercises

BMI > 35, which may interfere with ultrasonographic assessment

Non-compliance risk, such as irregular attendance or language barriers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic Floor Muscle Function Measured by Ultrasonography (mm displacement) | Baseline and Week 8
  Change in displacement of pelvic floor muscle during contraction, measured via transabdominal ultrasonography. Higher values indicate stronger muscle activity.
Female Sexual Function Index (FSFI) Total Score | Baseline and Week 8
  FSFI is a validated 19-item questionnaire (Score range: 2-36), with higher scores indicating better sexual function.
Heart Rate Variability (HRV) Index Measured with Elite HRV | Baseline and Week 8
  Time-domain and frequency-domain HRV parameters. Higher HRV indicates better autonomic balance.

SECONDARY OUTCOMES:
Pain Intensity During Intercourse Assessed by VAS (0-10 cm) | Baseline and Week 8
  VAS line score from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain.
Beck Anxiety Inventory (BAI) Total Score | Baseline and Week 8
  BAI includes 21 items scored 0-3 each (Total Score: 0-63); higher scores indicate worse anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Abdurrahim Yıldız, Assoc. Prof., Principal Investigator — Sakarya Applied Sciences University

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared after publication upon reasonable request.

REFERENCES:
- [Result] Nappi RE, Cucinella L, Martella S, Rossi M, Tiranini L, Martini E. Female sexual dysfunction (FSD): Prevalence and impact on quality of life (QoL). Maturitas. 2016 Dec;94:87-91. doi: 10.1016/j.maturitas.2016.09.013. Epub 2016 Sep 28. PMID 27823751
- [Result] Basson R, Wierman ME, van Lankveld J, Brotto L. Summary of the recommendations on sexual dysfunctions in women. J Sex Med. 2010 Jan;7(1 Pt 2):314-26. doi: 10.1111/j.1743-6109.2009.01617.x. PMID 20092441
- [Result] Bornstein J, Goldstein AT, Stockdale CK, Bergeron S, Pukall C, Zolnoun D, Coady D; consensus vulvar pain terminology committee of the International Society for the Study of Vulvovaginal Disease (ISSVD), the International Society for the Study of Women's Sexual Health (ISSWSH), and the International Pelvic Pain Society (IPPS). 2015 ISSVD, ISSWSH and IPPS Consensus Terminology and Classification of Persistent Vulvar Pain and Vulvodynia. Obstet Gynecol. 2016 Apr;127(4):745-751. doi: 10.1097/AOG.0000000000001359. PMID 27008217
- [Result] Buster JE. Managing female sexual dysfunction. Fertil Steril. 2013 Oct;100(4):905-15. doi: 10.1016/j.fertnstert.2013.08.026. PMID 24074537
- [Result] Berghmans B. Physiotherapy for pelvic pain and female sexual dysfunction: an untapped resource. Int Urogynecol J. 2018 May;29(5):631-638. doi: 10.1007/s00192-017-3536-8. Epub 2018 Jan 9. PMID 29318334
- [Result] Ege E, Akın B, Yaralı Arslan S, Bilgili N. (2010). Cinsel fonksiyon bozukluğu ve risk faktörleri. TÜBAV Bilim Dergisi, 3(2), 137-144.
- [Result] Oksuz E, Malhan S. Prevalence and risk factors for female sexual dysfunction in Turkish women. J Urol. 2006 Feb;175(2):654-8; discussion 658. doi: 10.1016/S0022-5347(05)00149-7. PMID 16407018
- [Result] Shifren JL, Monz BU, Russo PA, Segreti A, Johannes CB. Sexual problems and distress in United States women: prevalence and correlates. Obstet Gynecol. 2008 Nov;112(5):970-8. doi: 10.1097/AOG.0b013e3181898cdb. PMID 18978095